CLINICAL TRIAL: NCT04231175
Title: Dedicated MR Imaging vs Surgical Staging of Peritoneal Carcinomatosis in Colorectal Cancer Patients; a Multicenter Randomized Trial
Brief Title: Dedicated MR Imaging vs Surgical Staging of Peritoneal Carcinomatosis in Colorectal Cancer
Acronym: DISCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: M19DSC
Record Dates: First submitted 2019-10-31; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Colorectal Cancer; Peritoneal Carcinomatosis; MRI
Keywords: Colorectal cancer; Peritoneal Carcinomatosis; MRI; Randomization
MeSH Terms: conditions — Colorectal Neoplasms; Peritoneal Neoplasms

STUDY DESIGN:
Intervention Model Description: multi center randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental arm A (Experimental): patients will undergo dedicated MRI imaging of the pelvis, abdomen, and thorax. Based on the findings of the MRI scan patients will be allocated to one of the diagnostic/treatment options
  Interventions: Diagnostic Test: DWI MRI of the pelvis, abdomen and thorax
- arm B (No Intervention): patients will undergo the current standard diagnostic work-up of DLS at indication (MDT decision) and otherwise continue to CRS-HIPEC.

INTERVENTIONS:
Diagnostic Test: DWI MRI of the pelvis, abdomen and thorax — Patients in Arm A will receive a MRI scan of their pelvis, abdomen, and thorax before possible surgery. During the MRI standard Gadolinium contrast agent and Buscopan is intravenously administered, which is standard clinical practice in abdominal MR imaging. Total scan time is 35 minutes and includes T2 weighted, T1 weighted, Diffusion weighted and dynamic contrast enhanced imaging of the abdomen and the thorax. The findings of this scan will be used to determine whether to proceed with CRS/HIPEC, DLS and then possibly CRS-HIPEC, or palliative care.
  Arms: experimental arm A

SUMMARY:
MRI is a potentially powerful tool to reliably determine the intra-abdominal tumor load and relations with intra-abdominal organs. In recent years diffusion weighted MRI has proven its value as a highly sensitive technique to detect small malignant disease in a wide variety of cancers [1-3]. However, literature concerning the clinical impact of detecting peritoneal metastases with MRI is very limited. Therefore, there is a need for a large randomized multicenter trial to determine whether dedicated MRI can be used as a selection tool for CRS-HIPEC candidates in daily practice.

DETAILED DESCRIPTION:
HYPOTHESIS Staging with dedicated MRI will lead to a reduction of staging laparoscopies and explorative laparotomies in colorectal patients with PM to evaluate whether they may benefit from CRS-HIPEC

OBJECTIVES The goal is to perform a multicenter randomized study to compare a less invasive diagnostic workup ARM A (with MRI and surgical inspection reserved for borderline operable cases on MRI) to the standard diagnostic workup (ARM B, without MRI, with surgical staging to determine resectability based on a MDT decision) of patients with (suspected) peritoneal metastases. Surgical staging laparoscopies may largely be replaced by MRI (only reserved as a problem solver for borderline operable cases in ARM A). If it will be proven that MRI is an accurate, robust and cost-effective staging tool than this will result in a more patient friendly diagnostic workup with less futile surgical procedures.

STUDY DESIGN 4-year multicenter randomized controlled trial

STUDY POPULATION N=272 patients suspected of synchronous or metachronous peritoneal metastases of colorectal origin who are considered for CRS-HIPEC after CT imaging.

EXPERIMENTAL (ARM A) CRS-HIPEC candidates are selected based on MRI and only in borderline cases a surgical inspection will be performed

CONTROL (ARM B) Standard work-up including computed tomography and surgical inspection as appropriate (based on a MDT decision).

MAIN STUDY PARAMETERS/ENDPOINTS

Primary outcome:

Number of preventable unnecessary laparoscopies and explorative laparotomies.

NATURE AND EXTENT OF THE BURDEN AND RISKS ASSOCIATED WITH PARTICIPATION, BENEFIT AND GROUP RELATEDNESS:

MRI is a standard diagnostic procedure without the use of radiation. The MR sequences, MR-contrast agents and Buscopan (to minimize peristaltic bowel movements) are all commonly used in daily clinical practice. In addition, patients will be asked to drink 1L of pineapple juice 1-2 hours before the MRI (to minimize signal in the bowel lumen and optimize image quality), which is standard procedure in many clinics for MRCP and MR enterography. By acting upon the MRI findings in the experimental arm A, could result into new risks as oppose to standard clinical practice. However by introducing the borderline group ('yellow light' group) to receive diagnostic laparoscopy will minimize the possibility of over-staging a patient that would have received a successful CRS/HIPEC in de control arm. In our internal pilot data of 87 patients considered for CRS/HIPEC, no patients with a PCI of above 24 ended up receiving successful CRS/HIPEC and only 4 of the 15 patients that could have been assigned to the borderline group (were the trail to have run at that time) received successful CRS/HIPEC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspicion of colorectal peritoneal metastases and considered for CRS/HIPEC

  * Age ≥18 years
  * Written and signed informed consent
  * WHO 0-2
  * Able and willing to drink 1 liter of pineapple or blueberry juice

Exclusion Criteria:

* - Patients with contraindications for the MRI:
* Patients who have a heart pacemaker may not have an MRI scan
* Patients who have a metallic foreign body (metal sliver) in their body
* Patients with severe claustrophobia
* Ineligible to receive gadofosveset (Gadolinium) contrast (history of contrast allergy, impaired kidney function with a Glomerular Filtration Rate <30 ml/min/1.73m2)
* Ineligible to receive Buscopan
* Allergy for pineapple juice and blueberry juice.
* Patients with clinical contraindications for CRS/HIPEC
* Patients with radiological contra-indications for CRS/HIPEC observed on CT thorax/abdomen
* Massive mesenteric or small bowel involvement which would lead to short bowel syndrome if adequately resected
* Extra-peritoneal metastases for which CRS/HIPEC is not justifiable (such as lung metastases, skeletal metastases, and liver metastases)
* Inoperable retroperitoneal lymphadenopathy
* Patients with a known additional malignancy, unless o treated with curative intent at least five years ago. in situ cancers, basal cell carcinoma of the skin or squamous cell carcinoma of the skin that have undergone potentially curative therapy within the past five years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2023-10-28 (Estimated); Study Completion 2023-10-28 (Estimated)

PRIMARY OUTCOMES:
Number of preventable unnecessary laparoscopies and explorative laparotomies defined as: | 4 weeks
  (I) patients with a PCI<15 at laparoscopy or PCI>24 at laparotomy (II) incomplete CRS-HIPEC (R2A/R2B/open-close procedures)
Number of preventable unnecessary laparoscopies and explorative laparotomies defined as | 4 weeks
  (II) incomplete CRS-HIPEC (R2A/R2B/open-close procedures)

SECONDARY OUTCOMES:
- Number of additional extra-peritoneal findings | 4 weeks
  Number of additional extra-peritoneal findings
- Number of early recurrences (with-in 6 months after R1 resection and HIPEC) | 6 months
  - Number of early recurrences (with-in 6 months after R1 resection and HIPEC)
- Diagnostic performance of Peritoneal Cancer Index determined by MRI (MRI-PCI) to predict surgical Peritoneal Cancer Index (S-PCI). | 6 months
  - The Peritoneal Cancer Index (PCI) system reported by Sugerbaker [24] will be determined by indicating the presence of large (>5cm), moderate (<5cm - >0.5cm), small (<0.5cm) or no involvement in 13 abdominal regions
- Inter-observer agreement between different readers for DW-MRI. | 6 months
  Readers will evaluate the following MR criteria that might result in an incomplete CRS with a confidence level score (0 to 5):
  * MRI-PCI > 20
  * Extensive agglutinated intra-abdominal disease (stomach/liver/spleen/retrohepatic)
  * Extensive serosa involvement (>1.5 m bowel resection needed)
  * Extensive disease at diaphragmatic level (>1 cm in diameter)
  * Extensive extra-abdominal disease (>1 cm in diameter) in patients without neoadjuvant treatment
  * Presence and location of intra-abdominal enlarged lymph nodes
  * Ascites > 500 ml
  * Overall resectability based on MRI findings
Incremental cost-effectiveness ratio | 6 months
  The direct costs will include costs of standard treatment (chemotherapy and cytoreductive surgery), costs of diagnostic work-up (standard and MRI) and treatment of adverse events/surgical complications, follow-up visits, recurrences and palliative care (measured as possible within the trial period). From this the cost effectiveness will be determined.
Quality of Life between diagnostic arms by EORTC-C30 - | 6 months
  The following questionnaire will be used to measure HRQoL in patients EORTC-C30. This will be completed at baseline, 3 & 6 months following randomisation.
Quality of Life between diagnostic arms by EQ5D5L | 6 months
  The following questionnaire will be used to measure HRQoL in patients EQ5D5L. This will be completed at baseline, 3 & 6 months following

CONTACTS AND LOCATIONS:
Overall Officials: Max Lahaye, PhD MD, Principal Investigator — Antoni van Leeuwenhoek
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Engbersen MP, Rijsemus CJV, Nederend J, Aalbers AGJ, de Hingh IHJT, Retel V, Lambregts DMJ, Van der Hoeven EJRJ, Boerma D, Wiezer MJ, De Vries M, Madsen EVE, Brandt-Kerkhof ARM, Van Koeverden S, De Reuver PR, Beets-Tan RGH, Kok NFM, Lahaye MJ. Dedicated MRI staging versus surgical staging of peritoneal metastases in colorectal cancer patients considered for CRS-HIPEC; the DISCO randomized multicenter trial. BMC Cancer. 2021 Apr 26;21(1):464. doi: 10.1186/s12885-021-08168-x. PMID 33902498